CLINICAL TRIAL: NCT03146234
Title: Clinical Study of Redirected Autologous T Cells With a GPC3-targeted Chimeric Antigen Receptor in Patients With Refractory Hepatocellular Carcinoma
Brief Title: CAR-GPC3 T Cells in Patients With Refractory Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG1006
Record Dates: First submitted 2017-04-24; First posted 2017-05-09 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-GPC3 T cells (Experimental): Autologous T Cells with a GPC3-redirected Chimeric Antigen Receptor. Route of administration: Intravenous injection.
  Lymphodepletion conditioning regimen: A combination of fludarabine and cyclophosphamide will be administered at Day -6 to Day -3 prior to CAR-GPC3 T cells infusion.
  Interventions: Genetic: CAR-GPC3 T cells

INTERVENTIONS:
Genetic: CAR-GPC3 T cells — Self-controlled dose escalation will be applied to the first 3 - 6 subjects enrolled.
  Classical "3+3" dose escalation will be applied to subsequent subjects based on the self-controlled dose escalation study.
  Other Names: GPC3 Redirected Autologous Cells

SUMMARY:
This study is designed to determine the safety and efficacy of CAR-GPC3 T cells in patients with relapsed or refractory hepatocellular carcinoma. Single or multiple doses of GPC3-targeted CAR T cells will be given to subjects with unmet medical needs for which there are no effective therapies known at this time.

DETAILED DESCRIPTION:
A single arm, open-label pilot study is designed to determine the safety, tolerability and engraftment potential of CAR-GPC3 T cells in patients with GPC3-positive hepatocellular carcinoma.

Primary objectives:

Determine the safety, tolerability and cytokinetics of the autologous T cells transduced with the anti- GPC3 lentiviral vector in patients with hepatocellular carcinoma.

Secondary objectives:

Make a preliminary evaluation on the efficacy of CAR-GPC3 T cells in patients with hepatocellular carcinoma by the following parameters:

Objective response rate (ORR); Disease Control Rate (DCR); Time of tumor progression (TTP); Overall survival (OS).

ELIGIBILITY:
Inclusion criteria:

1. Age of 18-70 years;
2. Pathologically confirmed advanced hepatocellular carcinoma (HCC);
3. ≥1 measurable target lesion per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1);
4. Tumor tissue positive for GPC3 expression per immunohistochemical staining (IHC) assay;
5. Estimated survival > 12 weeks;
6. Child-Pugh grade A;
7. ECOG performance score of 0-1;
8. HBV-DNA < 200 IU/mL if positive for HBsAg or HBcAb. Patients positive for HBsAg shall receive anti-viral treatment per "The guideline of prevention and treatment for chronic hepatitis B: a 2015 update";
9. Have adequate venous access for apheresis or venous blood collection;
10. White blood cells ≥ 2.5 x 109/L, platelet ≥ 60×109/L, haemoglobin ≥ 9.0 g/dL, lymphocyte ≥ 0.4×109/L
11. Serum albumin ≥ 30 g/dL, serum lipase and amylase≤1.5 upper limit of normal (ULN), serum creatinine ≤ 1.5 ULN and endogenous creatinine clearance ≥ 40mL/min, ALT and AST ≤ 5 ULN, Serum total bilirubin ≤ 2.5 ULN, Prothrombin Time is less than 4s longer than normal;
12. Negative serum pregnancy test within 14 days before CAR T infusion, and with willingness to use reliable contraceptive methods to avoid pregnancy until 12 months after CAR T infusions for females of childbearing age; Having undergone sterilization procedure or with willingness to use reliable contraceptive methods to avoid pregnancy for males with female partner of childbearing age during the study;
13. Able to understand and sign the informed consent form

Exclusion criteria:

If the patient meets any of the exclusion criteria, the patient must be excluded from the study.

1. Pregnant or lactating female patients;
2. Positive serum tests for HCV, HIV, or syphilis;
3. Presence of HBV/HCV coinfection;
4. Presence of any uncontrollable active infection, such as, but not limited to, active tuberculosis
5. History of systemic administration of steroids (not including inhaled steroids), or other immunosuppressant drugs within 2 weeks before apheresis;
6. History of allergy to immunotherapy and related drugs, or β-lactam antibiotics, or history of other severe allergy;
7. History or current presence of hepatic encephalopathy;
8. Presence of ascites with clinical significance that is defined as positive focused physical examination for ascites, or ascites that requires treatment intervention (not including any ascites shown on image examinations without the need for clinical intervention);
9. ≥ 50% of normal liver occupied with HCC tumor tissue, or presence of tumor thrombus in the portal vein, or mesenteric vein, or inferior vena based on image analysis;
10. Presence of HCC metastatic lesion in the central nervous system, or presence of other diseases of central nervous system with clinical significance;
11. Presence of heart disease that requires treatment intervention, or poorly controlled hypertension (systolic pressure > 160 mmHg, or diastolic pressure > 100 mmHg);
12. Presence of active auto-immune disease that requires immunosuppressant treatment;
13. History of organ transplantation or currently on the waiting list for organ transplantation, including, but not limited to, liver transplantation;
14. Anti-HCC therapies including, but not limited to, surgical resection, interventional therapy, radiation therapy, chemotherapy, and immunotherapy, within 2 weeks before apheresis;
15. History of receiving anti-PD-1 or anti-PD-L1 monoclonal antibodies, or other immunotherapy;
16. History of other malignancies in the past 5 years, or presence of other active malignancies (not including cervical cancer in situ and basal cell carcinomas);
17. Presence of other serious diseases or conditions, including uncontrolled diabetes (HbA1c > 7% with treatment); severe cardiac dysfunction with LVEF < 45%; myocardial infarction, unstable angina, or unstable arrhythmia in the past 6 months pulmonary embolism; chronic obstructive pulmonary disease; interstitial lung disease; forced expiratory volume in 1 second (FEV1) < 60%, gastric ulcer; history of gastrointestinal bleeding, or confirmed tendency for gastrointestinal bleeding;
18. Determined by the investigator to be lack of compliance for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance | 24 weeks
  Study related adverse events are defined as signs above CTCAE Grade 3, laboratory toxicities and clinical events occurred at any time from the first day of infusion to week 24 that are "possibly", "likely", or "definitely" related to the study, including infusion related toxicity and CAR-GPC3 T cells related toxicity. Include but not limited to:
  Fever; Chills; Nausea, vomiting and other gastrointestinal symptoms; Fatigue; Hypotension; Respiratory distress; Tumor lysis syndrome; Cytokine release syndrome; Neutropenia, thrombocytopenia; Liver and kidney dysfunction; Other toxicities.

SECONDARY OUTCOMES:
Engraftment | 2 years
  Duration of in vivo survival of CAR-GPC3 T cells is defined as "engraftment". The primary engraftment endpoint is the number of DNA vector copies per mL blood of CAR-GPC3 T cells at regular intervals through week 4 following the initial infusion. Q-PCR for CAR-GPC3 vector sequences will be performed until any 2 sequential tests are negative, documented as engraftment and persistence of CAR-GPC3 T cells.

OTHER OUTCOMES:
Anti-tumor responses to CAR-GPC3 T cell infusions | 2 years
  Objective response rate (ORR); Progression-free survival (PFS); Time of tumor progression (TTP); Overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhai, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided